CLINICAL TRIAL: NCT05456451
Title: Investigation of the Effectiveness of Noninvasive Vagus Stimulation on Upper Extremity Functions in Parkinson's Disease
Brief Title: Effectiveness of Noninvasive Vagus Stimulation for Upper Extremity in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other); Acibadem Atakent University Hospital (Other); Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3616
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; Upper Extremity Dysfunction; Tremor
Keywords: vagus nerve stimulation; tremor; parkinson disease; upper extremity
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Intervention Model Description: The participants wit Parkinson disease, who has Hohen Yahr grade 2-3 will be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson group(pre and post treatment) (Experimental): 5 participants will be evaluated for tremor and autonomic dysfunction at pre and post treatment
  Interventions: Device: noninvasive vagus nerve srimulation

INTERVENTIONS:
Device: noninvasive vagus nerve srimulation — Non-invasive Vagus nerve stimulation (VNS) stimulates the vagus nerve through the ear via a headset. VNS is a non-pharmacological intervention with the potential to improve walking, cognition, fatigue, and autonomic functions in the treatment of Parkinson's disease.

SUMMARY:
Vagus nerve stimulation in the treatment of PD is a non-pharmacological intervention with the potential to improve gait, cognition, fatigue, and autonomic functions, but more evidence is needed for VSS in the treatment of PD. The potential mechanisms of VSS in the improvement seen in PD are explained by increased cholinergic transmission, decreased neuroinflammation, and enhanced NE release.

In this study, it was aimed to investigate the effects of non-invasive vagus nerve stimulation to be applied to patients with Parkinson's disease on tremor and vagus nerve activity in patients.

The tremor and autonomic activations of the participants will be evaluated at pre and post treatment.

DETAILED DESCRIPTION:
Vagus nerve stimulation in the treatment of PD is a non-pharmacological intervention with the potential to improve gait, cognition, fatigue, and autonomic functions, but more evidence is needed for VSS in the treatment of PD. The potential mechanisms of VSS in the improvement seen in PD are explained by increased cholinergic transmission, decreased neuroinflammation, and enhanced NE release.

5 patients who meet the inclusion criteria will be included in this prospectively planned study. As a vagus stimulation protocol, noninvasive auricular stimulation and stimulation frequency of 10 Hz, pulse width of 300 µs, biphasic application for 20 minutes will be applied to each patient 3 times on different days. Stimulations will be performed 3 times on 3 different days as the right ear, left ear and bilateral ear.

The tremor of the patients participating in the study will be evaluated with the smartphone application. After opening the phone application (G-Sensor), which is used to measure tremor, the patients will be asked to hold the phone in each hand at rest for 30 seconds and the tremor will be recorded. In this application, the maximum amplitude and frequency of the tremor in the 3D plane are calculated automatically.

The effect of vagus nerve stimulation on autonomic nervous system activity is evaluated using heart rate variability with Polar device.

The participants will be evaluated pre and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-65.
* Diagnosed with Parkinson's Disease by a specialist neurologist.
* Hoehn-Yahr stage 2-3.
* Having bilateral resting tremor of the hands.
* Being agreed to participate in the study.

Exclusion Criteria:

* Bilateral or unilateral previous injury to the vagus nerve (eg injury during carotid endarterectomy).
* Severe depression (Beck Depression Scale > 29)
* Current use of any other stimulation device, such as a pacemaker or other neurostimulator; current use of any other investigational device or drug.
* Medical or mental instability (diagnosis of personality disorder, psychosis, or substance abuse) that would prevent the subject from following the protocol timeline.
* Pregnancy or planning to become pregnant or breast-feed during the study period.
* Botox injections or any other upper extremity rehabilitation within 6 months prior to treatment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2022-09-25 (Estimated); Study Completion 2022-10-25 (Estimated)

PRIMARY OUTCOMES:
tremor | 1 day
  The tremor of the patients participating in the study will be evaluated with the smartphone application. After opening the phone application (G-Sensor), which is used to measure tremor, the patients will be asked to hold the phone in each hand at rest for 30 seconds and the tremor will be recorded. In this application, the maximum amplitude and frequency of the tremor in the 3D plane are calculated automatically. This application provides the opportunity to evaluate tremor numerically in patients with tremor, and there are studies where it has been used before in Parkinson's disease.
autonomic nervous system | 1 day
  The effect of vagus nerve stimulation on autonomic nervous system activity is evaluated using heart rate variability by using Polar device.

CONTACTS AND LOCATIONS:
Overall Officials: E. Efe Is, M.D., Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital; Ceyhun Basoglu, M.D., Principal Investigator — Acibadem Atakent University Hospital; Mustafa Corum, M.D., Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital; Ali Veysel Ozden, M.D., Principal Investigator — Bahçeşehir University
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
not decided